CLINICAL TRIAL: NCT06580470
Title: Improving Functioning Among Aging Women Veterans With Major Mental Illness
Brief Title: Improving Functioning Among Aging Women Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4792-W; RX004792 (Other Grant/Funding Number: VA Rehabilitation Research & Development)
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Menopause
Keywords: Menopause; Cognitive Behavioral Therapy; Veterans; Women's Health; Aging
MeSH Terms: interventions — Menopause

STUDY DESIGN:
Intervention Model Description: Cognitive Behavioral Therapy for Menopause (CBT-Meno) is an evidenced-based intervention that includes psychoeducation, cognitive, and behavioral strategies for coping with common menopause symptoms and experiences. In Aims 1 and 2, CBT-Meno materials and procedures will be tailored for women Veterans through an iterative process involving: a) data from preliminary studies and a pre-pilot trial; b) input from content area experts; and c) stakeholder advisory panels. This tailored version of CBT-Meno will then be tested in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tailored CBT-Meno (Experimental): Cognitive Behavioral Therapy for Menopause (CBT-Meno) is an evidenced-based intervention that includes psychoeducation, cognitive, and behavioral strategies for coping with common menopause symptoms and experiences. In Aims 1 and 2, CBT-Meno materials and procedures will be tailored for women Veterans through an iterative process involving: a) data from preliminary studies and a pre-pilot trial; b) input from content area experts; and c) stakeholder advisory panels. This tailored version of CBT-Meno will then be test in this clinical trial.
  Interventions: Behavioral: Tailored Cognitive Behavioral Therapy for Menopause

INTERVENTIONS:
Behavioral: Tailored Cognitive Behavioral Therapy for Menopause — Cognitive Behavioral Therapy for Menopause (CBT-Meno) is an evidenced-based intervention that includes psychoeducation, cognitive, and behavioral strategies for coping with common menopause symptoms and experiences. In Aims 1 and 2, CBT-Meno materials and procedures will be tailored for women Veterans through an iterative process involving: a) data from preliminary studies and a pre-pilot trial; b) input from content area experts; and c) stakeholder advisory panels. This tailored version of CBT-Meno will then be test in this clinical trial.
  Other Names: Tailored CBT-Meno

SUMMARY:
Women are the fastest-growing group of U.S. Veterans. Over half of those using VA care are 45 or older, with more age-related health concerns than civilian women. The VA urgently needs gender-informed strategies to ensure women Veterans receive tailored care that addresses their intersecting mental, physical, and age related health concerns, as well as gender-linked stressors. One prominent example is menopause, a health transition period that, for many women, can be associated with negative physical and mental health concerns that can worsen their functioning and quality of life. This project will: (1) integrate stakeholder feedback to tailor Cognitive Behavioral Therapy for Menopause (CBT-Meno) for women Veterans with menopause concerns; and (2) refine and evaluate tailored CBT-Meno as a treatment to address these intersecting needs in a clinical trial.

DETAILED DESCRIPTION:
Anticipated Impact on Veteran's Healthcare: The VA's commitment to serving all Veterans must include effective, gender-informed services that address the needs of women Veterans. This application will address this need by exploring one method of offering gender-informed care by tailoring an existing intervention to optimize functioning among mid-life and older women Veterans.

Background: Women are the fastest-growing cohort of Veterans. They have higher rates of age-related health concerns than non-Veteran women, experiences that are further complicated by intersecting mental, physical, and gender-linked stressors. One prominent example of this intersection is menopause, a health transition period that can be associated with negative health impacts and functional challenges. These difficulties can be further complicated for women Veterans given high rates of physical and mental health conditions as well as exposure to challenging experiences associated with military service (e.g., military sexual trauma, service connected conditions, combat exposure). The VA urgently needs interventions that integrate such knowledge to help VA healthcare providers effectively, respectfully, and efficiently address the needs of aging women Veterans via gender-informed, tailored approaches. Cognitive behavioral therapies for menopause (CBT-Meno) are promising treatments for disruptive menopause concerns, showing effectiveness among non-Veteran women for many menopause symptoms (i.e., sleep, hot flashes, anxiety, depression), and quality of life. However, CBT-Meno research has not addressed the needs and risk factors specific to women Veterans and is limited in assessing functional outcomes. Research and VA policy also highlight the need for gender-informed interventions to address women Veterans' health concerns, including menopause care.

Project Objectives: This proposed CDA-2 research study will address these clinical and research gaps by testing one approach for delivering gender-informed services to aging women Veterans by: (1) integrating stakeholder feedback to tailor Cognitive Behavioral Therapy for Menopause (CBT-Meno) for women Veterans with menopause concerns; and (2) refining and evaluating tailored CBT-Meno as a treatment to address the intersecting needs of women Veterans with menopause concerns. This application will first, develop a tailored version of CBT-Meno, to be delivered via telehealth, utilizing feedback from stakeholder panels to address the intersecting care needs of women Veterans with menopause concerns. Second, it will examine the initial acceptability of tailored CBT-Meno through a pre-pilot group with women Veterans with menopause concerns - seeking feedback from the women Veteran participants and the stakeholder panels to inform refinement of tailored CBT-Meno for testing in Aim 3. [Third, a single-arm pilot trial of tailored CBT-Meno will be conducted to examine the feasibility, acceptability and fidelity of tailored CBT-Meno, and its impact on women Veterans' functioning, quality of life, and menopause symptom severity among women Veterans 45 years with menopause concerns.

Project Methods: The tailoring of CBT-Meno will start with existing knowledge and incorporate input from stakeholder panels of women Veterans, VA providers, and women Veterans' healthcare leaders to create a first draft of tailored CBT-Meno, which will be used to examine its acceptability in a pre-pilot group with women Veterans aged 45 with menopause concerns (N=6). Next, findings will be integrated with additional stakeholder feedback to generate a finalized version of tailored CBT-Meno for testing in Aim 3. Then, tailored CBT-Meno will be tested in a single-arm pilot trial (N=48) enrolling the same population. Feasibility, acceptability, fidelity, and preliminary efficacy will be assessed via quantitative and qualitative methods. The trial will assess health, quality of life, and community functioning at Baseline, Post, and Follow-up timepoints.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* 45 years of age or older
* currently receiving services at the VA Maryland Healthcare System
* presence of at least one symptom rated "moderate" or above or two symptoms rated "mild" or above the Menopause Rating Scale (MRS)
* ability to participate in telehealth appointments

Exclusion Criteria:

* are engaging in moderate-to-severe substance use that would impact their ability to participate and/or would require a higher level of care (as determined by chart review)
* engagement in CBT-Meno, whether currently or in the past
* participated in Aim 1 as a Veteran stakeholder

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment, approximately 12 weeks
  To examine acceptability, the investigators will collect satisfaction ratings via the Client Satisfaction Questionnaire (CSQ-8) at post-treatment assessment. The CSQ-8 contains eight Likert scale items that ask about quality of service received and if services have been helpful and provides an overall score. Reliability/validity for the measure is good. The minimum score is 8 and the maximum score is 32, with greater scores indicating more client satisfaction.
Recruitment | At completion of study recruitment, approximately 1.5 years
  As a measure of feasibility, the investigators will evaluate recruitment by calculating the number of eligible participants (e.g., those that passed screening) divided by the number of potential participants that were approached for recruitment (# eligible ÷ # approached).
Retention Rate | Following completion of all intervention groups, approximately 2 years
  As a measure of feasibility, investigators will calculate retention rates defined as the percentage of enrolled participants who attend first 2 sessions ("engaged").
Outreach Efforts | Throughout intervention delivery, approximately 2 years
  As a measure of feasibility, investigators will examine our study outreach efforts by calculating the mean number of reminders and outreach contacts made for each participant during the course of treatment.
Suitability of Eligibility | At completion of study recruitment, approximately 1.5 years
  As a measure of feasibility, the investigators will evaluate suitability of eligibility criteria by calculating the number of participants enrolled in the study divided by the number eligible (e.g., those that passed screening;# enrolled ÷ # eligible).
Adherence rate | Following completion of all intervention groups, approximately 2 years
  As a measure of feasibility, investigators will calculate the adherence rate measured by treatment dropout percentages. This will be calculated as the number of participants who dropped out prior to completing treatment divided by the number who engaged (i.e., "engaged" = enrolled participants who attend first 2 sessions; #who dropped out prior to completing treatment ÷ # who engaged).

CONTACTS AND LOCATIONS:
Overall Officials: Haley Miles-McLean, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (2):
- United States (2):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Perry Point VA Medical Center VA Maryland Health Care System, Perry Point, MD, Perry Point, Maryland

IPD SHARING:
Plan to Share IPD: No